CLINICAL TRIAL: NCT03334396
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Baricitinib in Adult Patients With Moderate to Severe Atopic Dermatitis
Brief Title: A Study of Baricitinib (LY3009104) in Patients With Moderate to Severe Atopic Dermatitis
Acronym: BREEZE-AD1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16580; I4V-MC-JAHL (Other: Eli Lilly and Company); 2017-000870-12 (EudraCT Number)
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Results first posted 2020-01-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-01

CONDITIONS: Atopic Dermatitis
Keywords: eczema; atopic eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- 4 milligram (mg) Baricitinib (Experimental): 4 mg Baricitinib administered orally once daily. Placebo 1 mg and 2 mg administered orally every day to match.
  Interventions: Drug: Baricitinib; Drug: Placebo
- 2 mg Baricitinib (Experimental): 2 mg Baricitinib administered orally once daily. Placebo 1 mg and 4 mg administered orally every day to match.
  Interventions: Drug: Baricitinib; Drug: Placebo
- 1 mg Baricitinib (Experimental): 1 mg Baricitinib administered orally once daily. Placebo 2 mg and 4 mg administered orally every day to match.
  Interventions: Drug: Baricitinib; Drug: Placebo
- Placebo (Placebo Comparator): Placebo administered orally once daily.
  Interventions: Drug: Placebo
- 4 mg Baricitinib Maximum Extended Enrollment Cohort (Experimental): 4 mg Baricitinib administered orally once daily. Placebo 1 mg, and 2 mg administered orally every day to match.
  Interventions: Drug: Baricitinib; Drug: Placebo
- 2 mg Baricitinib Maximum Extended Enrollment Cohort (Experimental): 2 mg Baricitinib administered orally once daily. Placebo 1 mg and 4 mg administered orally every day to match.
  Interventions: Drug: Baricitinib; Drug: Placebo
- 1 mg Baricitinib Maximum Extended Enrollment Cohort (Experimental): 1 mg Baricitinib administered orally once daily. Placebo 2 mg and 4 mg administered orally every day to match.
  Interventions: Drug: Baricitinib; Drug: Placebo
- Placebo Maximum Extended Enrollment Cohort (Placebo Comparator): Placebo administered orally once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib — Administered orally.
  Other Names: LY3009104
  Arms: 1 mg Baricitinib; 1 mg Baricitinib Maximum Extended Enrollment Cohort; 2 mg Baricitinib; 2 mg Baricitinib Maximum Extended Enrollment Cohort; 4 mg Baricitinib Maximum Extended Enrollment Cohort; 4 milligram (mg) Baricitinib
Drug: Placebo — Administered orally.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of baricitinib as monotherapy in participants with moderate to severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with moderate to severe Atopic Dermatitis for at least 12 months.
* Have had inadequate response or intolerance to existing topical (applied to the skin) medications within 6 months preceding screening.
* Are willing to discontinue certain treatments for eczema (such as systemic and topical treatments during a washout period).
* Agree to use emollients daily.

Exclusion Criteria:

* Are currently experiencing or have a history of other concomitant skin conditions (e.g., psoriasis or lupus erythematosus), or a history of erythrodermic, refractory, or unstable skin disease that requires frequent hospitalizations and/or intravenous treatment for skin infections.
* A history of eczema herpeticum within 12 months, and/or a history of 2 or more episode of eczema herpeticum in the past.
* Participants who are currently experiencing a skin infection that requires treatment, or is currently being treated, with topical or systemic antibiotics.
* Have any serious illness that is anticipated to require the use of systemic corticosteroids or otherwise interfere with study participation or require active frequent monitoring (e.g., unstable chronic asthma).
* Have been treated with the following therapies:

  * Monoclonal antibody for less than 5 half-lives prior to randomization.
  * Received prior treatment with any oral Janus kinase (JAK) inhibitor.
  * Received any parenteral corticosteroids administered by intramuscular or intravenous (IV) injection within 2 weeks prior to study entry or within 6 weeks prior to planned randomization or are anticipated to require parenteral injection of corticosteroids during the study.
  * Have had an intra-articular corticosteroid injection within 2 weeks prior to study entry or within 6 weeks prior to planned randomization.
* Have high blood pressure characterized by a repeated systolic blood pressure >160 millimeters of mercury (mm Hg) or diastolic blood pressure >100 mm Hg.
* Have had major surgery within the past eight weeks or are planning major surgery during the study.
* Have experienced any of the following within 12 weeks of screening: venous thromboembolic event (VTE), myocardial infarction (MI), unstable ischemic heart disease, stroke, or New York Heart Association Stage III/IV heart failure.
* Have a history of recurrent (≥ 2) VTE or are considered at high risk of VTE as deemed by the investigator.
* Have a history or presence of cardiovascular, respiratory, hepatic, chronic liver disease gastrointestinal, endocrine, hematological, neurological, lymphoproliferative disease or neuropsychiatric disorders or any other serious and/or unstable illness.
* Have a current or recent clinically serious viral, bacterial, fungal, or parasitic infection including herpes zoster, tuberculosis.
* Have specific laboratory abnormalities.
* Have received certain treatments that are contraindicated.
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2019-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (93):
- Czechia (9):
  - Kozni ambulance Kutna Hora, s.r.o., Kutná Hora, Central Bohemia
  - Clintrial, s.r.o., Prague, Hl. M. Praha
  - Fakultni nemocnice Kralovske Vinohrady, Prague, Hl. M. Praha
  - Fakultni Nemocnice v Motole, Prague, Hl. M. Praha
  - Nemocnice Na Bulovce, Prague, Hl. M. Praha
  - Nemocnice Novy Jicin a.s., Nový Jičín, Moravskoslezský kraj
  - Fakultni Nemocnice Plzen, Plzen, Jizni Predmesti, Plzeň Region
  - Fakultni Nemocnice U svate Anny, Brno, South Moravian
  - Krajska zdravotni a.s. - Masarykova nemocnice v Usti nad Labem, o.z., Ústí nad Labem, Ustecký Kraj
- Aarhus Universitehospital Marselisborg Centret, Aarhus, Denmark
- France (8):
  - Hopital Saint-Louis, Paris, Cedex 10
  - CHU de Bordeaux Hopital Saint Andre, Bordeaux
  - CHRU de Brest - Hôpital Morvan, Brest
  - CHU Grenoble Alpes, Grenoble Cédex 9
  - Chru De Nantes Hotel-Dieu, Nantes
  - CHU de Nice Hopital de L'Archet, Nice
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hopital Larrey, Toulouse
- Germany (21):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Klinikum der Universität München, München, Bavaria
  - Gemeinschaftspraxis Mahlow, Blankenfelde-Mahlow, Brandenburg
  - Rosenpark Research Geschäftsbereich der Rosenparkklinik GmbH, Darmstadt, Hesse
  - Klinikum der Johann Wolfgang Goethe-Universität Frankfurt, Frankfurt am Main, Hesse
  - Dermatologisches Zentrum Osnabrück Nord, Bramsche, Lower Saxony
  - Universitätsmedizin Göttingen, Göttingen, Lower Saxony
  - Universitätsmedizin Rostock, Rostock, Mecklenburg-Vorpommern
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Praxis Dr. Thomas Dirschka, Wuppertal, North Rhine-Westphalia
  - Praxis Gerlach, Dresden, Saxony
  - Universitätsklinikum Carl Gustav Carus, Dresden, Saxony
  - Universität Leipzig - Universitätsklinikum, Leipzig, Saxony
  - Universitätsklinikum Otto-von-Guericke-Universität, Magdeburg, Saxony-Anhalt
  - Hautarztzentrum Kiel, Kiel, Schleswig-Holstein
  - Universitätsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein
  - Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - Rothhaar Studien GmbH, Berlin
  - ISA GmbH, Berlin
  - Praxis für Ganzheitliche Dermatologie im Ärztehaus, Berlin
  - TFS Trial Form Support GmbH, Hamburg
- India (12):
  - King George Hospital, Vizag, Andhra Pradesh
  - Panchshil Hospital, Ahmedabad, Gujarat
  - Byramjee Jeejeebhoy Medical College & Civil Hospital, Ahmedabad, Gujarat
  - M S Ramaiah Medical College Hospital, Bangalore, Karnataka
  - Dr. D. Y. Patil Medical College & Hospital, Navi Mumbai, Maharashtra
  - Jehangir Hospital, Pune, Maharashtra
  - Seth GS Medical College & KEM Hospital, Mumbai, Maharshtra
  - All India Institue of Medical Sciences (AIIMS), New Delhi, National Capital Territory of Delhi
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Chennai Meenakshi Multispeciality Hospital, Chennai, Tamil Nadu
  - Gandhi Hospital, Secunderabad, Telangana
  - MV Hospital and Research Centre, Lucknow, Uttar Pradesh
- Italy (5):
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliera - Universitaria Pisana, Pisa
  - Policlinico di Tor Vergata, Roma
  - Ospedale Policlinico Giambattista Rossi, Borgo Roma, Verona
- Japan (16):
  - Kawashima Dermatology Clinic, Ichikawa-shi, Chiba
  - Fumimori Clinic, Fukuoka, Fukuoka
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Queen's Square Dermatology and Allergology, Nishi-ku, Yokohama-city, Kanagawa
  - Yokohama City Minato Red Cross Hospital, Yokohama, Kanagawa
  - Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Kume Clinic, Nishi-ku Sakai-shi, Osaka
  - Shimane University Hospital, Izumo, Shimane
  - JA Shizuoka Kohseiren Enshu Hospital, Hamamatsu, Shizuoka
  - Iidabashi Clinic, Chiyoda-ku, Tokyo
  - Nihonbashi Sakura Clinic, Chuo-ku, Tokyo
  - Sumire Dermatology Clinic, Edogawa-ku, Tokyo
  - NTT Medical Center Tokyo, Shinagawa-KU, Tokyo
  - Shirasaki Clinic, Takaoka-shi, Toyama
  - Yamanashi Prefectural Central Hospital, Kofu, Yamanashi
  - Fukuoka University Hospital, Fukuoka
- Mexico (8):
  - Grupo Médico CAMINO S.C., Mexico City, Mexico City
  - Hospital de Jesus I.A.P., Mexico City, Mexico City
  - Clínica Enfermedades Crónicas y Procedimientos Especiales SC, Morella, Michoacán
  - CRI Centro Regiomontano de Investigacion S.C., Monterrey, Nuevo León
  - Hospital Univ. Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - JM Research S.C., Cuernavaca
  - RM Pharma Specialists S.A. de C.V., Distrito Federal
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C, Durango
- Russia (6):
  - GBUZ Clinical dermatology and venereological dispensary, Krasnodar
  - State scientific centre for dermatovenerology and cosmetolog, Moscow
  - Russian state medical-stomatological university n.a. Evdokimov, Moscow
  - SPb SBHI Skin-venerologic dispensary #10, Saint Petersburg
  - LLC ArsVitae NorthWest, Saint Petersburg
  - LLC Medical Center "Kurator", Saint Petersburg
- Taiwan (7):
  - Chang Gung Memorial Hospital - Kaohsiung, Kaohsiung City
  - Taipei Medical University- Shuang Ho Hospital, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital - Taipei, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Katoh N, Takita Y, Isaka Y, Nishikawa A, Torisu-Itakura H, Saeki H. Pooled Safety Analysis of Baricitinib in Adult Participants with Atopic Dermatitis in the Japanese Subpopulation from Six Randomized Clinical Trials. Dermatol Ther (Heidelb). 2022 Dec;12(12):2765-2779. doi: 10.1007/s13555-022-00828-5. Epub 2022 Oct 18. PMID 36255569
- [Derived] Silverberg JI, DeLozier A, Sun L, Thyssen JP, Kim B, Yosipovitch G, Nunes FP, Gugiu PC, Doll HA, Eichenfield LF. Psychometric properties of the itch numeric rating scale, skin pain numeric rating scale, and atopic dermatitis sleep scale in adult patients with moderate-to-severe atopic dermatitis. Health Qual Life Outcomes. 2021 Oct 23;19(1):247. doi: 10.1186/s12955-021-01877-8. PMID 34688290
- [Derived] Thyssen JP, Buhl T, Fernandez-Penas P, Kabashima K, Chen S, Lu N, DeLozier AM, Casillas M, Stander S. Baricitinib Rapidly Improves Skin Pain Resulting in Improved Quality of Life for Patients with Atopic Dermatitis: Analyses from BREEZE-AD1, 2, and 7. Dermatol Ther (Heidelb). 2021 Oct;11(5):1599-1611. doi: 10.1007/s13555-021-00577-x. Epub 2021 Jul 18. PMID 34275122
- [Derived] King B, Maari C, Lain E, Silverberg JI, Issa M, Holzwarth K, Brinker D, Cardillo T, Nunes FP, Simpson EL. Extended Safety Analysis of Baricitinib 2 mg in Adult Patients with Atopic Dermatitis: An Integrated Analysis from Eight Randomized Clinical Trials. Am J Clin Dermatol. 2021 May;22(3):395-405. doi: 10.1007/s40257-021-00602-x. Epub 2021 Apr 7. PMID 33826132
- [Derived] Reich K, DeLozier AM, Nunes FP, Thyssen JP, Eichenfield LF, Wollenberg A, Ross Terres JA, Watts SD, Chen YF, Simpson EL, Silverberg JI. Baricitinib improves symptoms in patients with moderate-to-severe atopic dermatitis and inadequate response to topical corticosteroids: patient-reported outcomes from two randomized monotherapy phase III trials. J Dermatolog Treat. 2022 May;33(3):1521-1530. doi: 10.1080/09546634.2020.1839008. Epub 2020 Nov 22. PMID 33222559
- See also: A Study of Baricitinib (LY3009104) in Adults With Moderate to Severe Atopic Dermatitis (Eczema) (BREEZE-AD1) — https://www.lillytrialguide.com/en-US/studies/eczema/JAHL#?postal=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed double blind treatment phase had option to enter extension study I4V-MC-JAHN (NCT03334435).
Groups:
- 1 mg Baricitinib; 1 mg Baricitinib MEE: 1 mg Baricitinib administered orally once daily.
- 2 mg Baricitinib; 2 mg Baricitinib MEE: 2 mg Baricitinib administered orally once daily.
- 4 mg Baricitinib; 4 mg Baricitinib MEE: 4 mg Baricitinib administered orally once daily.
- Placebo Maximum Extended Enrollment (MEE): Placebo administered orally once daily.
Period: Overall Study
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib | Placebo Maximum Extended Enrollment (MEE) | 1 mg Baricitinib MEE | 2 mg Baricitinib MEE | 4 mg Baricitinib MEE
Started | 249 | 127 | 123 | 125 | 15 | 5 | 8 | 8
Received at Least One Dose of Study Drug | 249 | 127 | 123 | 125 | 15 | 5 | 8 | 8
Completed | 226 | 116 | 113 | 120 | 12 | 4 | 5 | 7
Not Completed | 23 | 11 | 10 | 5 | 3 | 1 | 3 | 1
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 10 | 4 | 1 | 3 | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 10 | 5 | 7 | 2 | 2 | 1 | 2 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Ineligible | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Started New Job | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants. Results for maximum extended enrollment (MEE) participants will be reported within 1-year after the study completion.
Groups:
- 1 mg Baricitinib MEE: 1 mg Baricitinib administered orally once daily. .
- Total: Total of all reporting groups
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib | Placebo Maximum Extended Enrollment (MEE) | 1 mg Baricitinib MEE | 2 mg Baricitinib MEE | 4 mg Baricitinib MEE | Total
Number analyzed (Participants) | 249 | 127 | 123 | 125 | 15 | 5 | 8 | 8 | 660
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Between 18 and 65 years | 242 | 127 | 118 | 121 | 15 | 5 | 6 | 8 | 642
  >=65 years | 7 | 0 | 5 | 4 | 0 | 0 | 1 | 0 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 49 | 41 | 42 | 6 | 2 | 0 | 2 | 243
  Male | 148 | 78 | 82 | 83 | 9 | 3 | 8 | 6 | 417
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 14 | 7 | 7 | 2 | 0 | 0 | 0 | 0 | 30
  Asian | 73 | 40 | 35 | 41 | 15 | 5 | 8 | 8 | 225
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
  White | 147 | 74 | 75 | 70 | 0 | 0 | 0 | 0 | 366
  More than one race | 13 | 6 | 5 | 10 | 0 | 0 | 0 | 0 | 34
  Unknown or Not Reported | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Czechia | 36 | 11 | 11 | 18 | 0 | 0 | 0 | 0 | 76
  Japan | 45 | 23 | 21 | 22 | 0 | 0 | 0 | 0 | 111
  Taiwan | 25 | 13 | 13 | 12 | 0 | 0 | 0 | 0 | 63
  Italy | 17 | 8 | 6 | 13 | 0 | 0 | 0 | 0 | 44
  Mexico | 32 | 15 | 17 | 9 | 0 | 0 | 0 | 0 | 73
  France | 15 | 4 | 13 | 7 | 0 | 0 | 0 | 0 | 39
  Germany | 67 | 44 | 37 | 30 | 0 | 0 | 0 | 0 | 178
  India | 1 | 2 | 1 | 6 | 15 | 5 | 8 | 8 | 46
  Russia | 11 | 7 | 4 | 8 | 0 | 0 | 0 | 0 | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Investigator's Global Assessment (IGA) of 0 or 1 With a ≥ 2 Point Improvement (Placebo, 2 mg, or 4 mg Baricitinib)
Description: The IGA measures the investigator's global assessment of the participant's overall severity of their atopic dermatitis (AD), based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification.
Time Frame: 16 Weeks
Population: All participants randomized to placebo, 2 mg, or 4 mg of study drug. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (MEE) arms/groups but only for the main global study arms/groups.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 249 | 123 | 125
percentage of participants | 4.8 | 11.4 | 16.8
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.020, Regression, Logistic; Odds Ratio (OR) = 2.61, 95% CI 2-sided [1.17 to 5.84]
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.10, 95% CI 2-sided [1.93 to 8.70]

2. Secondary Outcome: Percentage of Participants Achieving IGA of 0 or 1 With a ≥ 2 Point Improvement (Placebo, 1 mg Baricitinib)
Description: The IGA measures the investigator's global assessment of the participant's overall severity of their AD, based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification.
Time Frame: 16 Weeks
Population: All participants randomized to placebo or 1 mg of study drug. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (MEE) arms/groups but only for the main global study arms/groups.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib
Number analyzed (Participants) | 249 | 127
percentage of participants | 4.8 | 11.8
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.014, Regression, Logistic; Odds Ratio (OR) = 2.72, 95% CI 2-sided [1.23 to 6.01]

3. Secondary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index 75 (EASI75)
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe). The EASI75 is defined as a ≥ 75% improvement from baseline in the EASI score.
Time Frame: 16 Weeks
Population: All randomized participants. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (MEE) arms/groups but only for the main global study arms/groups.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 249 | 127 | 123 | 125
percentage of participants | 8.8 | 17.3 | 18.7 | 24.8
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.032, Regression, Logistic; Odds Ratio (OR) = 2.03, 95% CI 2-sided [1.06 to 3.88]
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 2.46, 95% CI 2-sided [1.29 to 4.67]
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.72, 95% CI 2-sided [2.01 to 6.89]

4. Secondary Outcome: Percentage of Participants Achieving EASI90
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe). The EASI90 is defined as a ≥ 90% improvement from baseline in the EASI score.
Time Frame: 16 Weeks
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 249 | 127 | 123 | 125
percentage of participants | 4.8 | 8.7 | 10.6 | 16.0
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.210, Regression, Logistic; Odds Ratio (OR) = 1.73, 95% CI 2-sided [0.74 to 4.05]
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.029, Regression, Logistic; Odds Ratio (OR) = 2.50, 95% CI 2-sided [1.10 to 5.70]
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.13, 95% CI 2-sided [1.91 to 8.91]

5. Secondary Outcome: Percent Change From Baseline in EASI Score
Description: The EASI assesses objective physician estimates of 2 dimensions of AD - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe).
  Least Square (LS) Means were calculated using a MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effect
Time Frame: Baseline, 16 Weeks
Population: All randomized participants who had Week 16 EASI data. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (MEE) arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 71 | 52 | 52 | 70
percent change | -34.82 (3.64) | -48.22 (4.52) | -51.89 (4.29) | -59.36 (3.84)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.021, Mixed Models Analysis; Mean Difference (Final Values) = -13.40, 95% CI 2-sided [-24.77 to -2.03], Standard Error of Mean 5.78
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = -17.07, 95% CI 2-sided [-28.05 to -6.10], Standard Error of Mean 5.57
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -24.54, 95% CI 2-sided [-34.84 to -14.24], Standard Error of Mean 5.23

6. Secondary Outcome: Percentage of Participants Achieving SCORing Atopic Dermatitis 75 (SCORAD75)
Description: The SCORAD index uses the rule of nines to assess disease extent and evaluates 6 clinical characteristics to determine disease severity: (1) erythema, (2) edema/papulation, (3) oozing/crusts, (4) excoriation, (5) lichenification, and (6) dryness on a scale of 0 to 3 (0=absence, 1=mild, 2=moderate, 3=severe). The SCORAD index also assesses subjective symptoms of pruritus and sleep loss with visual analog scale (VAS) where 0 is no itching or no trouble sleeping and 10 is unbearable itching or a lot of trouble sleeping. These 3 aspects: extent of disease (A: 0-1-2), disease severity (B: 0-18), & subjective symptoms (C: 0-20) combine using A/5 + 7*B/2+ C to give a maximum possible score of 103, where 0 = no disease and 103 = severe disease. The SCORAD75 responder is defined as a participant who achieves a ≥ 75% improvement from baseline in the SCORAD score.
Time Frame: 16 Weeks
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 249 | 127 | 123 | 125
percentage of participants | 1.2 | 5.5 | 7.3 | 10.4
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.025, Regression, Logistic; Odds Ratio (OR) = 4.28, 95% CI 2-sided [1.20 to 15.24]
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.004, Regression, Logistic; Odds Ratio (OR) = 6.14, 95% CI 2-sided [1.79 to 20.99]
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 8.76, 95% CI 2-sided [2.68 to 28.58]

7. Secondary Outcome: Percentage of Participants Achieving a 4-Point Improvement in Itch Numeric Rating Scale (NRS)
Description: The Itch Numeric Rating Scale (NRS) is a participant-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no itch" and 10 representing "worst itch imaginable." Overall severity of a participants itching is indicated by selecting the number, using a daily diary, that best describes the worst level of itching in the past 24 hours.
Time Frame: 16 Weeks
Population: All randomized participants with a Baseline Itch NRS score >=4. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (MEE) arms/groups but only for the main global study arms/groups.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 222 | 105 | 100 | 107
percentage of participants | 7.2 | 10.5 | 12.0 | 21.5
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.246, Regression, Logistic; Odds Ratio (OR) = 1.60, 95% CI 2-sided [0.72 to 3.56]
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.169, Regression, Logistic; Odds Ratio (OR) = 1.73, 95% CI 2-sided [0.79 to 3.77]
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.62, 95% CI 2-sided [1.82 to 7.18]

8. Secondary Outcome: Change From Baseline in the Score of Item 2 of the Atopic Dermatitis Sleep Scale (ADSS)
Description: Atopic Dermatitis Sleep Scale (ADSS) is a 3-item, participant-administered questionnaire developed to assess the impact of itch on sleep including difficulty falling asleep, frequency of waking, and difficulty getting back to sleep last night. Item 2, frequency of waking last night is reported by selecting the number of times they woke up each night, ranging from 0 to 29 times,where the higher a number indicates a worse outcome. The ADSS is designed to be completed daily, using a daily diary, with respondents thinking about sleep "last night." Each item is scored individually.
  LS Means were calculated using a MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by- visit-interaction as fixed continuous effects.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants with Week 16 ADSS Item 2 (frequency of waking) data. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (MEE) arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 68 | 52 | 50 | 68
units on a scale | -0.84 (0.15) | -1.21 (0.18) | -1.04 (0.17) | -1.42 (0.16)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.103, Mixed Models Analysis; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.82 to 0.08]
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.352, Mixed Models Analysis; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.65 to 0.23]
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.006, Mixed Models Analysis; Mean Difference (Final Values) = -0.58, 95% CI 2-sided [-1.00 to -0.17]

9. Secondary Outcome: Change From Baseline in the Skin Pain Numeric Rating Scale (NRS)
Description: Skin Pain NRS is a participant-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no pain" and 10 representing "worst pain imaginable." Overall severity of a participant's skin pain is indicated by selecting the number, using a daily diary, that best describes the worst level of skin pain in the past 24 hours.
  LS Means were calculated using a MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants with Week 16 Skin Pain NRS data. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (MEE) arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 68 | 52 | 50 | 68
units on a scale | -0.84 (0.24) | -1.92 (0.30) | -1.58 (0.29) | -1.93 (0.26)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.005, Mixed Models Analysis; Mean Difference (Final Values) = -1.08, 95% CI 2-sided [-1.84 to -0.32]
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.051, Mixed Models Analysis; Mean Difference (Final Values) = -0.74, 95% CI 2-sided [-1.48 to 0.00]
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = -1.09, 95% CI 2-sided [-1.79 to -0.39]

10. Secondary Outcome: Percentage of Participants Achieving EASI50
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100%) and the severity of 4 clinical signs (erythema, edema/papulation, excoriation, and lichenification) each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head and neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2 and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe). The EASI50 is defined as a ≥ 50% improvement from baseline in EASI score.
Time Frame: 16 Weeks
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 249 | 127 | 123 | 125
percentage of participants | 15.3 | 26.0 | 30.1 | 41.6
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.019, Regression, Logistic; Odds Ratio (OR) = 1.90, 95% CI 2-sided [1.11 to 3.25]
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Mean Difference (Final Values) = 2.44, 95% CI 2-sided [1.44 to 4.14]
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Mean Difference (Final Values) = 4.18, 95% CI 2-sided [2.51 to 6.96]

11. Secondary Outcome: Percentage of Participants Achieving IGA of 0
Description: as for outcome 2
Time Frame: 16 Weeks
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 249 | 127 | 123 | 125
percentage of participants | 0.8 | 1.6 | 2.4 | 1.6
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.424, Regression, Logistic; Odds Ratio (OR) = 1.98, 95% CI 2-sided [0.37 to 10.63]
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.182, Regression, Logistic; Odds Ratio (OR) = 2.89, 95% CI 2-sided [0.61 to 13.75]
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.441, Regression, Logistic; Odds Ratio (OR) = 1.94, 95% CI 2-sided [0.36 to 10.41]

12. Secondary Outcome: Change From Baseline in SCORAD
Description: The SCORAD index uses the rule of nines to assess disease extent and evaluates 6 clinical characteristics to determine disease severity: (1) erythema, (2) edema/papulation, (3) oozing/crusts, (4) excoriation, (5) lichenification, and (6) dryness on a scale of 0 to 3 (0=absence, 1=mild, 2=moderate, 3=severe). The SCORAD index also assesses subjective symptoms of pruritus and sleep loss with VAS where 0 is no itching or no trouble sleeping and 10 is unbearable itching or a lot of trouble sleeping. These 3 aspects: extent of disease (A: 0-1-2), disease severity (B: 0-18), & subjective symptoms (C: 0-20) combine using A/5 + 7*B/2+ C to give a maximum possible score of 103, where 0 = no disease and 103 = severe disease.
  LS Means were calculated using a MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants with Week 16 SCORAD data. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (MEE) arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 71 | 52 | 52 | 70
units on a scale | -13.51 (2.00) | -18.85 (2.48) | -21.47 (2.36) | -28.30 (2.10)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.093, Mixed Models Analysis; Mean Difference (Final Values) = -5.34, 95% CI 2-sided [-11.57 to 0.90], Standard Error of Mean 3.17
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.010, Mixed Models Analysis; Mean Difference (Final Values) = -7.97, 95% CI 2-sided [-14.01 to -1.92], Standard Error of Mean 3.07
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -14.79, 95% CI 2-sided [-20.46 to -9.13], Standard Error of Mean 2.88

13. Secondary Outcome: Percentage of Participants Achieving SCORAD90
Description: The SCORAD index uses the rule of nines to assess disease extent and evaluates 6 clinical characteristics to determine disease severity: (1) erythema, (2) edema/papulation, (3) oozing/crusts, (4) excoriation, (5) lichenification, and (6) dryness on a scale of 0 to 3 (0=absence, 1=mild, 2=moderate, 3=severe). The SCORAD index also assesses subjective symptoms of pruritus and sleep loss with VAS where 0 is no itching or no trouble sleeping and 10 is unbearable itching or a lot of trouble sleeping. These 3 aspects: extent of disease (A: 0-1-2), disease severity (B: 0-18), & subjective symptoms (C: 0-20) combine using A/5 + 7*B/2+ C to give a maximum possible score of 103, where 0 = no disease and 103 = severe disease. SCORAD90 is defined as a ≥ 90% improvement from baseline in the SCORAD score.
Time Frame: 16 Weeks
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 249 | 127 | 123 | 125
percentage of participants | 0.8 | 0.8 | 2.4 | 2.4
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.874, Regression, Logistic; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.17 to 7.77]
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.176, Regression, Logistic; Odds Ratio (OR) = 2.88, 95% CI 2-sided [0.62 to 13.36]
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.201, Regression, Logistic; Odds Ratio (OR) = 2.72, 95% CI 2-sided [0.59 to 12.65]

14. Secondary Outcome: Change From Baseline in Body Surface Area (BSA) Affected
Description: Body surface area affected by AD will be assessed for 4 separate body regions and is collected as part of the EASI assessment: head and neck, trunk (including genital region), upper extremities, and lower extremities (including the buttocks). Each body region will be assessed for disease extent ranging from 0% to 100% involvement. The overall total percentage will be reported based off of all 4 body regions combined, after applying specific multipliers to the different body regions to account for the percent of the total BSA represented by each of the 4 regions. Use the percentage of skin affected for each region (0 to 100%) in EASI as follows: BSA Total = 0.1*BSAhead and neck + 0.3*BSAtrunk + 0.2* BSAupper limbs + 0.4*BSAlower limbs.
  LS Means were calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants with Week 16 BSA data. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (MEE) arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 71 | 52 | 52 | 70
units on a scale | -14.80 (1.82) | -20.79 (2.26) | -20.14 (2.16) | -25.96 (1.93)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.039, Mixed Models Analysis; Mean Difference (Final Values) = -5.99, 95% CI 2-sided [-11.67 to -0.31], Standard Error of Mean 2.88
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.058, Mixed Models Analysis; Mean Difference (Final Values) = -5.34, 95% CI 2-sided [-10.86 to 0.18], Standard Error of Mean 2.80
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -11.16, 95% CI 2-sided [-16.33 to -5.98], Standard Deviation 2.63

15. Secondary Outcome: Percentage of Participants Developing Skin Infections Requiring Antibiotic Treatment
Description: Percentage of participants developing skin infections requiring antibiotic treatment.
Time Frame: 16 Weeks
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 249 | 127 | 123 | 125
percentage of participants | 4.4 | 0.8 | 4.9 | 3.2
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.067, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.799, Fisher Exact
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.782, Fisher Exact

16. Secondary Outcome: Percent Change From Baseline in Itch NRS
Description: The Itch NRS is a participant-administered, 11-point horizontal scale, with 0 representing "no itch" and 10 representing "worst itch imaginable." Overall severity of a participant's itching is indicated by selecting the number, using a daily diary, that best describes the worst level of itching in the past 24 hours.
  LS Means were calculated using a MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants with Week 16 Itch NRS data. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (MEE) arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 68 | 52 | 50 | 68
Percent Change | -12.04 (4.65) | -31.30 (5.70) | -29.43 (5.45) | -36.55 (4.88)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.009, Mixed Models Analysis; Mean Difference (Final Values) = -19.25, 95% CI 2-sided [-33.69 to -4.81], Standard Error of Mean 7.33
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.015, Mixed Models Analysis; Mean Difference (Final Values) = -17.39, 95% CI 2-sided [-31.43 to -3.35], Standard Error of Mean 7.13
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -24.50, 95% CI 2-sided [-37.71 to -11.30], Standard Error of Mean 6.71

17. Secondary Outcome: Change From Baseline in the Total Score of the Patient Oriented Eczema Measure (POEM)
Description: The POEM is a 7-item self-assessment questionnaire that assesses disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) on a scale ranging from 0-4 (0 = no days, 1 = 1-2 days, 2 = 3-4 days, 3 = 5-6 days, 4 = everyday). The sum of the 7 items gives the total POEM score of 0 (absent disease) to 28 (severe disease). High scores are indicative of more severe disease and poor quality of life.
  LS Means were calculated using a MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants with Week 16 POEM data. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (MEE) arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 72 | 53 | 52 | 70
units on a scale | -2.68 (0.76) | -5.32 (0.93) | -6.26 (0.91) | -7.84 (0.80)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.028, Mixed Models Analysis; Mean Difference (Final Values) = -2.63, 95% CI 2-sided [-4.98 to -0.29], Standard Error of Mean 1.19
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = -3.58, 95% CI 2-sided [-5.89 to -1.27], Standard Error of Mean 1.17
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -5.16, 95% CI 2-sided [-7.33 to -2.99], Standard Error of Mean 1.10

18. Secondary Outcome: Change From Baseline in the Patient Global Impression of Severity-Atopic Dermatitis (PGI-S-AD) Score
Description: The PGI-S-AD asked the participant to evaluate the severity of the disease at that point in time on a single-item, 5-point scale, using a daily diary. The same category labels used in the Physician's Global Assessment were used for the PGI-S-AD, i.e., "(0) no symptoms", "(1) very mild", "(2) mild" "(3) moderate", and "(4) severe."
  LS Means were calculated using a MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants with Week 16 PGI-S-AD data. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (MEE) arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 68 | 52 | 50 | 68
units on a scale | -0.31 (0.09) | -0.58 (0.12) | -0.58 (0.11) | -0.77 (0.10)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.069, Mixed Models Analysis; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-0.56 to 0.02], Standard Error of Mean 0.15
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.066, Mixed Models Analysis; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-0.56 to 0.02], Standard Error of Mean 0.15
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-0.73 to -0.19], Standard Error of Mean 0.14

19. Secondary Outcome: Change From Baseline on the Hospital Anxiety and Depression Scale (HADS)
Description: The HADS is a participant-rated instrument used to assess both anxiety and depression. This instrument consists of 14 item questionnaire, each item is rated on a 4-point scale, giving maximum scores of 21 for anxiety and depression. Scores of 11 or more on either subscale are considered to be a significant 'case' of psychological morbidity, while scores of 8-10 represent 'borderline' and 0-7, 'normal.' LS Means were calculated using a MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants with Week 16 HADS data. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (MEE) arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 71 | 51 | 52 | 70
units on a scale
  Anxiety | -0.90 (0.28) | -1.35 (0.34) | -1.83 (0.33) | -2.05 (0.30)
  Depression | -0.37 (0.27) | -1.04 (0.34) | -1.40 (0.32) | -1.50 (0.29)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; HADS Anxiety; Test type: Superiority; p = 0.305, Mixed Models Analysis; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-1.30 to 0.41], Standard Error of Mean 0.43
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; HADS Anxiety; Test type: Superiority; p = 0.029, Mixed Models Analysis; Mean Difference (Final Values) = -0.93, 95% CI 2-sided [-1.77 to -0.10], Standard Error of Mean 0.42
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; HADS Anxiety; Test type: Superiority; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = -1.15, 95% CI 2-sided [-1.93 to -0.36], Standard Error of Mean 0.40
Statistical Analysis 4: Comparison: Placebo vs 1 mg Baricitinib; HADS Depression; Test type: Superiority; p = 0.113, Mixed Models Analysis; Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-1.51 to 0.16], Standard Error of Mean 0.43
Statistical Analysis 5: Comparison: Placebo vs 2 mg Baricitinib; HADS Depression; Test type: Superiority; p = 0.014, Mixed Models Analysis; Mean Difference (Final Values) = -1.03, 95% CI 2-sided [-1.85 to -0.22], Standard Error of Mean 0.42
Statistical Analysis 6: Comparison: Placebo vs 4 mg Baricitinib; HADS Depression; Test type: Superiority; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = -1.14, 95% CI 2-sided [-1.91 to -0.37], Standard Error of Mean 0.39

20. Secondary Outcome: Change From Baseline in the Dermatology Life Quality Index (DLQI)
Description: The DLQI is a simple, participant-administered,10 question, validated, quality-of-life questionnaire that covers 6 domains including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. The recall period of this scale is over the last "week." Response categories include "not at all," "a lot," and "very much," with corresponding scores of 1, 2, and 3, respectively, and at unanswered ("not relevant") responses scored as "0." Scores range from 0 to 30 (less to more impairment), and a 4-point change from baseline is considered as the minimal clinically important difference threshold.
  LS Means were calculated using a MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants with Week 16 DLQI data. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (MEE) arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 71 | 52 | 52 | 70
units on a scale | -2.46 (0.57) | -4.64 (0.70) | -4.30 (0.68) | -6.76 (0.60)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.015, Mixed Models Analysis; Mean Difference (Final Values) = -2.17, 95% CI 2-sided [-3.92 to -0.42], Standard Error of Mean 0.89
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.036, Mixed Models Analysis; Mean Difference (Final Values) = -1.84, 95% CI 2-sided [-3.56 to -0.12], Standard Error of Mean 0.87
Statistical Analysis 3: Comparison: Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -4.30, 95% CI 2-sided [-5.91 to -2.69], Standard Error of Mean 0.82

21. Secondary Outcome: Change From Baseline on the Work Productivity and Activity Impairment - Atopic Dermatitis (WPAI-AD) Questionnaire
Description: The WPAI-AD participant questionnaire was developed to measure the effect of general health and symptom severity on work productivity and regular activities in the 7 days prior to the visit. The WPAI-AD consists of 6 items grouped in 4 domains: absenteeism (work time missed), presenteeism (impairment at work/reduced on-the-job effectiveness), work productivity loss (overall work impairment/absenteeism plus presenteeism), and activity impairment, that range from 0% to 100%, with higher values indicating greater impairment.
  LS Means were calculated using a MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants with Week 16 WPAI-AD data. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (MEE) arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 70 | 51 | 52 | 70
units on a scale
  Absenteeism: number analyzed (Participants) | 48 | 30 | 27 | 40
  Absenteeism | -0.49 (1.68) | -4.54 (2.15) | -0.84 (2.23) | -3.89 (1.88)
  Presenteeism: number analyzed (Participants) | 48 | 30 | 27 | 39
  Presenteeism | -2.89 (2.60) | -9.75 (3.37) | -11.53 (3.44) | -15.17 (2.95)
  Work Productivity Loss: number analyzed (Participants) | 48 | 30 | 27 | 39
  Work Productivity Loss | -2.57 (2.89) | -11.23 (3.75) | -9.06 (3.83) | -13.85 (3.29)
  Activity Impairment | -5.67 (2.16) | -12.98 (2.63) | -10.80 (2.57) | -22.20 (2.30)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Percentage of Absenteeism Change from Baseline; Test type: Superiority; p = 0.136, Mixed Models Analysis; Mean Difference (Final Values) = -4.05, 95% CI 2-sided [-9.39 to 1.29], Standard Error of Mean 2.70
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Percentage of Absenteeism Change from Baseline; Test type: Superiority; p = 0.898, Mixed Models Analysis; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-5.81 to 5.10], Standard Error of Mean 2.76
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Percentage of Absenteeism Change from Baseline; Test type: Superiority; p = 0.174, Mixed Models Analysis; Mean Difference (Final Values) = -3.40, 95% CI 2-sided [-8.32 to 1.52], Standard Error of Mean 2.49
Statistical Analysis 4: Comparison: Placebo vs 1 mg Baricitinib; Percentage of Presenteeism (Reduced Productivity While at Work) Change from Baseline; Test type: Superiority; p = 0.104, Mixed Models Analysis; Mean Difference (Final Values) = -6.86, 95% CI 2-sided [-15.13 to 1.41], Standard Error of Mean 4.19
Statistical Analysis 5: Comparison: Placebo vs 2 mg Baricitinib; Percentage of Presenteeism (Reduced Productivity While at Work) Change from Baseline; Test type: Superiority; p = 0.045, Mixed Models Analysis; Mean Difference (Final Values) = -8.64, 95% CI 2-sided [-17.09 to -0.19], Standard Error of Mean 4.28
Statistical Analysis 6: Comparison: Placebo vs 4 mg Baricitinib; Percentage of Presenteeism (Reduced Productivity While at Work) Change from Baseline; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = -12.28, 95% CI 2-sided [-19.97 to -4.59], Standard Error of Mean 3.90
Statistical Analysis 7: Comparison: Placebo vs 1 mg Baricitinib; Work Productivity Loss (Percentage Overall Work Impairment/Absenteeism Plus Presenteeism) Change from Baseline; Test type: Superiority; p = 0.066, Mixed Models Analysis; Mean Difference (Final Values) = -8.66, 95% CI 2-sided [-17.89 to 0.57], Standard Error of Mean 4.67
Statistical Analysis 8: Comparison: Placebo vs 2 mg Baricitinib; Work Productivity Loss (Percentage Overall Work Impairment/Absenteeism Plus Presenteeism) Change from Baseline; Test type: Superiority; p = 0.175, Mixed Models Analysis; Mean Difference (Final Values) = -6.49, 95% CI 2-sided [-15.89 to 2.91], Standard Error of Mean 4.76
Statistical Analysis 9: Comparison: Placebo vs 4 mg Baricitinib; Work Productivity Loss (Percentage Overall Work Impairment/Absenteeism Plus Presenteeism) Change from Baseline; Test type: Superiority; p = 0.010, Mixed Models Analysis; Mean Difference (Final Values) = -11.28, 95% CI 2-sided [-19.84 to -2.72], Standard Error of Mean 4.34
Statistical Analysis 10: Comparison: Placebo vs 1 mg Baricitinib; Percentage of Activity Impairment Change from Baseline; Test type: Superiority; p = 0.030, Mixed Models Analysis; Mean Difference (Final Values) = -7.31, 95% CI 2-sided [-13.93 to -0.70], Standard Error of Mean 3.36
Statistical Analysis 11: Comparison: Placebo vs 2 mg Baricitinib; Percentage of Activity Impairment Change from Baseline; Test type: Superiority; p = 0.122, Mixed Models Analysis; Mean Difference (Final Values) = -5.13, 95% CI 2-sided [-11.65 to 1.39], Standard Error of Mean 3.31
Statistical Analysis 12: Comparison: Placebo vs 4 mg Baricitinib; Percentage of Activity Impairment Change from Baseline; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -16.52, 95% CI 2-sided [-22.64 to -10.41], Standard Error of Mean 3.11

22. Secondary Outcome: Change From Baseline on the European Quality of Life-5 Dimensions 5 Levels (EQ-5D-5L) Index Score United States and United Kingdom Algorithm
Description: EQ-5D-5L is a 2-part measurement. The first part is comprised of the following 5 participant-reported dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses are used to derive the health state index scores using the United Kingdom (UK) algorithm, with scores ranging from -0.594 to 1, and the United States (US) algorithm, with scores ranging from -0.109 to 1, with higher score indicating better health state.
  LS Means were calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants with Week 16 EQ-5D-5L Health State Index US and UK data. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (MEE) arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 70 | 51 | 52 | 70
units on a scale
  Health State Index Score (US Algorithm) | 0.01 (0.01) | 0.05 (0.02) | 0.05 (0.02) | 0.09 (0.01)
  Health State Index Score (UK Algorithm) | 0.01 (0.02) | 0.07 (0.02) | 0.07 (0.02) | 0.13 (0.02)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Health State Index Score (US algorithm); Test type: Superiority; p = 0.061, Mixed Models Analysis; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.00 to 0.08], Standard Error of Mean 0.02
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Health State Index Score (US algorithm); Test type: Superiority; p = 0.060, Mixed Models Analysis; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.00 to 0.08], Standard Error of Mean 0.02
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Health State Index Score (US algorithm); Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [0.04 to 0.12], Standard Error of Mean 0.02
Statistical Analysis 4: Comparison: Placebo vs 1 mg Baricitinib; Health State Index Score (UK Algorithm); Test type: Superiority; p = 0.046, Mixed Models Analysis; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [0.00 to 0.11], Standard Error of Mean 0.03
Statistical Analysis 5: Comparison: Placebo vs 2 mg Baricitinib; Health State Index Score (UK Algorithm); Test type: Superiority; p = 0.059, Mixed Models Analysis; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.00 to 0.11], Standard Error of Mean 0.03
Statistical Analysis 6: Comparison: Placebo vs 4 mg Baricitinib; Health State Index Score (UK algorithm); Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [0.06 to 0.16], Standard Error of Mean 0.03

23. Secondary Outcome: Change From Baseline on the European Quality of Life-5 Dimensions 5 Levels (EQ-5D-5L) Visual Analog Score (VAS)
Description: EQ-5D-5L is a 2-part measurement. The second part is assessed using a visual analog scale (VAS) that ranged from 0 to 100 millimeter (mm), where 0 is the worst health you can imagine and 100 is the best health you can imagine.
  LS Means were calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants with Week 16 EQ-5D-5L VAS data. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (MEE) arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: millimeters
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 70 | 51 | 52 | 70
millimeters | 2.00 (2.04) | 4.97 (2.53) | 3.35 (2.41) | 9.05 (2.17)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; EQ-5D-5L VAS Score; Test type: Superiority; p = 0.356, Mixed Models Analysis; Mean Difference (Final Values) = 2.97, 95% CI 2-sided [-3.36 to 9.30], Standard Error of Mean 3.21
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; EQ-5D-5L VAS Score; Test type: Superiority; p = 0.668, Mixed Models Analysis; Mean Difference (Final Values) = 1.34, 95% CI 2-sided [-4.81 to 7.50], Standard Error of Mean 3.13
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; EQ-5D-5L VAS Score; Test type: Superiority; p = 0.017, Mixed Models Analysis; Mean Difference (Final Values) = 7.05, 95% CI 2-sided [1.25 to 12.86], Standard Error of Mean 2.95

24. Secondary Outcome: Percentage of Participants Achieving Investigator's Global Assessment (IGA) of 0 or 1 With a ≥ 2 Point Improvement
Description: as for outcome 2
Time Frame: 4 Weeks
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 249 | 127 | 123 | 125
percentage of participants | 2.4 | 3.1 | 8.9 | 10.4
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.603, Regression, Logistic; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.41 to 4.71]
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 4.08, 95% CI 2-sided [1.50 to 11.12]
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 4.72, 95% CI 2-sided [1.78 to 12.55]

ADVERSE EVENTS:
Time Frame: Baseline Up to 20 weeks
Description: All randomized participants who received at least one dose of study drug.
Groups:
- Placebo Maximum Extended Enrollment: Placebo administered orally once daily.
- 1 mg Baricitinib Maximum Extended Enrollment: 1 mg Baricitinib administered orally once daily.
- 2 mg Baricitinib Maximum Extended Enrollment: 2 mg Baricitinib administered orally once daily.
- 4 mg Baricitinib Maximum Extended Enrollment: 4 mg Baricitinib administered orally once daily.
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib | Placebo Maximum Extended Enrollment | 1 mg Baricitinib Maximum Extended Enrollment | 2 mg Baricitinib Maximum Extended Enrollment | 4 mg Baricitinib Maximum Extended Enrollment
All-Cause Mortality (participants affected / at risk) | 0/249 | 0/127 | 0/123 | 0/125 | 0/15 | 0/5 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 6/249 | 1/127 | 0/123 | 2/125 | 0/15 | 0/5 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 55/249 | 37/127 | 34/123 | 29/125 | 3/15 | 1/5 | 2/8 | 3/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=249) | 1 mg Baricitinib (N=127) | 2 mg Baricitinib (N=123) | 4 mg Baricitinib (N=125) | Placebo Maximum Extended Enrollment (N=15) | 1 mg Baricitinib Maximum Extended Enrollment (N=5) | 2 mg Baricitinib Maximum Extended Enrollment (N=8) | 4 mg Baricitinib Maximum Extended Enrollment (N=8)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=249) | 1 mg Baricitinib (N=127) | 2 mg Baricitinib (N=123) | 4 mg Baricitinib (N=125) | Placebo Maximum Extended Enrollment (N=15) | 1 mg Baricitinib Maximum Extended Enrollment (N=5) | 2 mg Baricitinib Maximum Extended Enrollment (N=8) | 4 mg Baricitinib Maximum Extended Enrollment (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 7 (8) | 9 (9) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 26 (28) | 22 (25) | 12 (14) | 12 (17) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 3 (4) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Urinary tract infection (Infections and infestations) | 4 (4) | 1 (1) | 2 (2) | 4 (7) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 1/101 (1) | 0/49 (0) | 0/41 (0) | 0/42 (0) | 1/6 (1) | 0/2 (0) | 0/0 (0) | 0/2 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 16 (17) | 7 (8) | 14 (15) | 10 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT03334396/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-16): https://cdn.clinicaltrials.gov/large-docs/96/NCT03334396/SAP_001.pdf